CLINICAL TRIAL: NCT02861456
Title: Feasibility of Using Functional Progression to Guide the Treatment of Adolescent Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Selhorst, Physical Therapist/Principle Investigator, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB16-00032
Record Dates: First submitted 2016-08-03; First posted 2016-08-10 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Low Back Pain; Spondylolysis; Spondylolisthesis
Keywords: Adolescent; Low Back Pain; Athlete
MeSH Terms: conditions — Low Back Pain; Spondylolysis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care Group (Active Comparator): Patient in the treatment arm will receive the Standard Model of Care as prescribed for their condition by their physician including but not limited to Advanced imaging, Rest, Bracing, Physical Therapy, and Medication.
  Interventions: Other: Standard Model of Care
- Functional Progression Group (Experimental): Patients who are randomized to the alternative model of care to guide treatment will not have advanced imaging done and will be referred directly to physical therapy care . If the patient is able to functional progress through phase I and II of physical therapy within 3 weeks and phase III within 5 weeks then they return to sport. If patient are unable to progress the are put on rest as a presumed vertebral injury (spondylolysis).
  Interventions: Other: Alternative Model of Care

INTERVENTIONS:
Other: Standard Model of Care
  Arms: Standard Care Group
Other: Alternative Model of Care
  Other Names: Functional progression program
  Arms: Functional Progression Group

SUMMARY:
The goal of the proposed research is to test the feasibility of a functional progression program to reduce cost and possible radiation exposure for adolescent athletes with low back pain. Specifically the investigators plan to test the feasibility of using progression in rehabilitation to pragmatically differentially diagnose and treat adolescent athletes with low back pain, instead of using advanced imaging which is the current practice. The investigators propose to recruit 20 participants, with 10 of usual care (advanced imaging) and 10 of proposed intervention (functional progression) to assess the feasibility of using functional progress to guide treatment. The outcomes measured will be number of days for rest, time to start regular rehabilitation, pain experienced, functional outcomes, ability to return to sport, time needed to return to sport. If this pilot demonstrates the feasibility and a decreased rate of advanced imaging and similar clinical outcomes the investigators plan to progress this work into larger trials.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common complaint in adolescent athletes, with rates reported as high as 50% by the mid-teen years. Although low back pain in adolescent athletes may result from several different pathologies, spondylolysis--a fracture at the pars interarticularis--is the most common cause in this demographic, with a prevalence as high as 47%. The recommended treatment of spondylolysis and non-specific mechanical LBP is quite different. Patients with mechanical LBP are recommended to stay active, and perform rehabilitation if necessary, while the primary treatment for spondylolysis is rest for 3 months, physical therapy and bracing as needed. With the diagnosis of spondylolysis being fairly common in young athletes with low back pain, physicians need to have a high index of suspicion in making the diagnosis. Advanced imaging is often necessary to confidently rule in or out the diagnosis of spondylolysis. Advanced imaging increases diagnostic accuracy, but adds to the cost and potentially considerable radiation exposure. However, advanced imaging may not be necessary to effectively treat adolescents with low back pain.

Function, not imaging, is used to determine when a patient has healed from a spondylolytic injury. In fact, results of healing on imaging have no association with clinical outcome. Most defects do not heal with non-operative treatment suggesting that a successful clinical outcome does not depend on healing of the lesion. The functional progress that patients make is markedly different between patients with mechanical LBP and patients with a spondylolysis. The majority of adolescents with mechanical LBP can make a full functional recovery on their own or with a short period of rehabilitation. A patient with a spondylolytic injury may demonstrate an inability to make a full return to activity with rehabilitation and requires a period of rest from sport and high level activity to make a full functional recovery. Due to the differences in progression between mechanical LBP and spondylolysis, functional progress could be used to differentially diagnose these conditions. If effective, using functional progress instead of advanced imaging would be more cost-effective and expose the patient to significantly less radiation. In a retrospective review of adolescent patients presenting to the investigators sports medicine clinic with LBP, 80% had advanced imaging performed due to a concern of spondylolysis. Thirty-two percent of patients were positive for spondylolysis on advanced imaging, and 11% of patients had multiple advanced imaging performed due to lack of progress. No other significant findings were noted on advanced imaging. By using functional progress to determine the course of care, and only using advanced imaging when a patient does not respond to conservative care, there is the potential to significantly reduce the need for advanced imaging.

The primary risk of using functional progress in physical therapy (PT) instead of advanced imaging to determine to the course of care in adolescents with LBP is a delayed diagnosis for those who fail to respond to conservative care. The risk of missing a sinister pathology mimicking LBP can be minimized with a thorough clinical evaluation and radiographs if warranted. The results of the investigators' previous work demonstrate that early PT care in patients with a spondylolytic injury is safe and reduces time to return to sport. In a retrospective review with a cross-sectional follow-up, patients with an acute spondylolysis who began physical therapy as soon a 4 weeks (mean of 2 months) made a quicker functional recovery back to all activity and had similar clinical outcomes at 1-5 year follow-ups. A delayed diagnosis does not negatively impact long-term functional outcomes for patients with a spondylolysis as duration of symptoms is not found to be associated with outcome. Using logistic regression on the same dataset as above to determine factors associated with good short and long-term clinical outcomes, duration of symtpoms or time to diagnosis was not found to impact outcomes. On the other hand, delaying PT care to obtain advanced imaging is found to negatively impact outcomes in patients with mechanical LBP.

This project will lay the groundwork to demonstrate the feasibility of a functional progression to treat adolescent athletes with LBP. If successful, additional study will be proposed to test the effectiveness of intervention (functional progression) as compared to usual care (imaging) in improving the recovery outcome of LBP. Ultimately, this research would lead to change in the way adolescent athletes with LBP are treated, resulting in decreased cost, decreased exposure to radiation, and decreased time to begin rehabilitation. The results of this work would positively impact patients, clinicians, and decreased the costs to the health care system.

Control Cohort A series of 10 individuals who meet the inclusion criteria and are patients of the sports medicine physicians (Dr.s James MacDonald, Ravindran), physicians who are not recruiting patients for the experimental cohort but are still co-investigators, will serve as a non-randomized control cohort of typical clinical care and outcomes.

Description of the functional progression to guide treatment protocol. (Figure 1) Patients will be evaluated by their physician to determine appropriateness for participation in this study. Patients who meet the inclusion criteria and consent to participate in the pilot study as a part of the experimental cohort will not have advanced imaging done and will be referred directly to PT care for 2 times per week for 3 weeks. The functional progression protocol will be performed by physical therapists trained in the treatment and progression protocol. Patients will perform phase I of the PT protocol and progress to phase II as able without an increase in pain and with sufficiently proper mechanics. (Table 1) Patients will be assessed at each session to determine if they meet the criteria to begin the next step of functional PT progression back to sport. (Table 2) Those patients who meet these criteria within the designated 3 week period will progress into the next phase of functional PT for return to sport activity with an additional 2 weeks of PT. If these patients progress well in this third phase, and are able to meet the return to sport criteria, they will be discharged from PT and monitored by phone for recurrence of symptoms until 2 months. (Table 3) Those patients who do not progress through phase I or II functionally or without pain will be braced, as determined by their physician, and placed on rest from all activities excepting ADL's and their PT home exercise program and will be treated as patients with a presumed spondylolysis. Additionally, patients who are unable to meet the return to sport criteria within 5 weeks of PT will be braced, as deemed necessary by their physician, and placed on rest from all activities except ADL's and their PT home exercise program and will be treated as having a presumed spondylolysis. These patients will follow care appropriate for the condition. They will rest from sport until >2 months after initial evaluation , be braced as necessary, and ultimately complete 4 weeks of PT care to progress them as able back to sport activity. Patients who are treated as having a presumed spondylolysis will not be returned to sport before 3 months of rest as this period of rest has been found to produce optimal results.(El Rassi et al., 2013) Patients will have monthly re-evaluations with their physician until discharge. If at any point the patient is not responding as expected or the physician has concerns over the patient's safety, the physician can take the appropriate steps they feel are necessary for the safety of the patient. Patients who are classified as non-responders will be those who do not progress as expected for the typical course of mechanical LBP or spondylolysis.

Specific Outcome Variables

1. Advanced imaging use during the episode of care: Computed tomography (CT), single-photon emission computed tomography (SPECT), and magnetic resonance imaging (MRI).
2. Total cost will be calculated as the billed costs of physician visits, physical therapy visits, radiographs, advanced imaging, prescribed brace, and prescribed medication.
3. Total number of PT visits will be calculated as the number of physical therapy visits completed for the LBP episode of care.
4. The number of days from when the physician initially evaluates the patient and places them on hold from sport activity to when the patient was cleared to return to sport.
5. , Clinical outcomes: Modified Odom's Criteria, and Micheli Functional Scale. Ability to return to sport This pilot study will not be randomized. All patients consenting to participate will be treated according to the treatment approach the co-investigating physicians have agreed to perform.

Blinding No blinding will be performed in this pilot trial as it is not feasible to blind either the clinicians or the patient to the treatment cohort.

Data Analysis Descriptive statistics of the patient demographics and outcome variables will be reported. The two treatment groups will be compared based on cost, imaging usage, and outcomes but will not perform statistical analysis due to the small sample size.

Treatment received Patient Characteristics (eg gender, age) Injury characteristics (eg duration of symptoms, type of symptoms Number of patients utilizing advanced imaging. Total cost of episode of care for LBP Total number of PT visits. Number of days to return to all sporting activity Clinical outcomes (eg pain, function, patient perceived improvement)

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-19 years old
2. Primary complaint of acute low back pain (<3months)
3. Participates in some type of athletic activity on a regular basis (>2 times a week)
4. Pain increases with lumbar extension

Exclusion Criteria:

1. Advanced imaging performed already (MRI, SPECT, CT)
2. Red flags present (bowel/bladder problems, saddle anesthesia, progressive neurological deficits, recent fever or infection, unexplained weight loss, unable to change symptoms with mechanical testing)
3. Numbness and tingling in any lumbar dermatome
4. Previous rest from sport >4 weeks without improved symptoms
5. Other orthopedic injury or condition that would alter the plan of care for LBP (i.e. pregnancy, concomitant anterior cruciate ligament tear)
6. History of lumbar surgery

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Utilization of advanced imaging | Approximately 3 months (Discharge from medical care (both physician and physical therapist))
  Advanced imaging will be defined as anything beyond radiography (x-ray) used to diagnose patients low back pain
Total cost of care | Approximately 3 months (Discharge from medical care (both physician and physical therapist))
  Total billed from hospital for the low back pain episode of care

SECONDARY OUTCOMES:
The number of days to return to all sporting activity. | Approximately 3 months (Discharge from medical care (both physician and physical therapist))
  The total number of days from when the patient begins the study to the date when they are released to return to sport by the health care provider
Change in Numeric Pain Rating Scale | Baseline, Approximately 3 months (Discharge from medical care (both physician and physical therapist))
  The Numeric Pain rating scale asks the patient their highest pain in the last 24 hours. The Numeric Pain Rating Scale is a 0-10 scale subjectively assessing a patients perceived level of pain. With 0 on the scale = to no pain, and 10 = to the worst pain imaginable.
Change in Micheli Functional Scale | Baseline, Approximately 3 months (Discharge from medical care (both physician and physical therapist))
  The Micheli Functional Scale is a self-reported measure of functional ability and pain on a 0-100 scale with 0 being no disability and 100 representing maximum disability. This scale has been found to have validity and reliability in young athletes with LBP.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Selhorst, DPT, Principal Investigator — Nationwide Children's Hospital
Locations (4):
- United States (4):
  - Nationwide Children's Hospital Sports and Ortho PT East Broad, Columbus, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT Dublin, Dublin, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT New Albany, New Albany, Ohio
  - Nationwide Children's Hospital Sports and Orthopedic PT Westerville location, Westerville, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balague F, Dutoit G, Waldburger M. Low back pain in schoolchildren. An epidemiological study. Scand J Rehabil Med. 1988;20(4):175-9. PMID 2976526
- [Background] Burton AK, Clarke RD, McClune TD, Tillotson KM. The natural history of low back pain in adolescents. Spine (Phila Pa 1976). 1996 Oct 15;21(20):2323-8. doi: 10.1097/00007632-199610150-00004. PMID 8915066
- [Background] Ebrall PS. The epidemiology of male adolescent low back pain in a north suburban population of Melbourne, Australia. J Manipulative Physiol Ther. 1994 Sep;17(7):447-53. PMID 7989878
- [Background] Micheli LJ, Wood R. Back pain in young athletes. Significant differences from adults in causes and patterns. Arch Pediatr Adolesc Med. 1995 Jan;149(1):15-8. doi: 10.1001/archpedi.1995.02170130017004. PMID 7827653
- [Background] d'Hemecourt PA, Zurakowski D, d'Hemecourt CA, Curtis C, Ugrinow V, Deriu L, Micheli LJ. Validation of a new instrument for evaluating low back pain in the young athlete. Clin J Sport Med. 2012 May;22(3):244-8. doi: 10.1097/JSM.0b013e318249a3ce. PMID 22382433
- [Background] Miller R, Beck NA, Sampson NR, Zhu X, Flynn JM, Drummond D. Imaging modalities for low back pain in children: a review of spondyloysis and undiagnosed mechanical back pain. J Pediatr Orthop. 2013 Apr-May;33(3):282-8. doi: 10.1097/BPO.0b013e318287fffb. PMID 23482264
- [Background] El Rassi G, Takemitsu M, Glutting J, Shah SA. Effect of sports modification on clinical outcome in children and adolescent athletes with symptomatic lumbar spondylolysis. Am J Phys Med Rehabil. 2013 Dec;92(12):1070-4. doi: 10.1097/PHM.0b013e318296da7e. PMID 24141103
- [Background] Iwamoto J, Sato Y, Takeda T, Matsumoto H. Return to sports activity by athletes after treatment of spondylolysis. World J Orthop. 2010 Nov 18;1(1):26-30. doi: 10.5312/wjo.v1.i1.26. PMID 22474624 (Retraction: PMID 29564215 World J Orthop. 2018 Mar 18;9(3):58-59)
- [Background] Selhorst M, Fischer A, Graft K, Ravindran R, Peters E, Rodenberg R, Welder E, MacDonald J. Timing of Physical Therapy Referral in Adolescent Athletes With Acute Spondylolysis: A Retrospective Chart Review. Clin J Sport Med. 2017 May;27(3):296-301. doi: 10.1097/JSM.0000000000000334. PMID 27347866
- [Background] Klein G, Mehlman CT, McCarty M. Nonoperative treatment of spondylolysis and grade I spondylolisthesis in children and young adults: a meta-analysis of observational studies. J Pediatr Orthop. 2009 Mar;29(2):146-56. doi: 10.1097/BPO.0b013e3181977fc5. PMID 19352240
- [Background] Congeni J, McCulloch J, Swanson K. Lumbar spondylolysis. A study of natural progression in athletes. Am J Sports Med. 1997 Mar-Apr;25(2):248-53. doi: 10.1177/036354659702500220. PMID 9079183
- [Background] Iwamoto J, Takeda T, Wakano K. Returning athletes with severe low back pain and spondylolysis to original sporting activities with conservative treatment. Scand J Med Sci Sports. 2004 Dec;14(6):346-51. doi: 10.1111/j.1600-0838.2004.00379.x. PMID 15546329
- [Background] Childs JD, Fritz JM, Wu SS, Flynn TW, Wainner RS, Robertson EK, Kim FS, George SZ. Implications of early and guideline adherent physical therapy for low back pain on utilization and costs. BMC Health Serv Res. 2015 Apr 9;15:150. doi: 10.1186/s12913-015-0830-3. PMID 25880898